CLINICAL TRIAL: NCT00608322
Title: Randomized Double-blind Placebo-controlled Trial of Inhaled Nitric Oxide for the Treatment of Microcirculatory Dysfunction and Organ Failure in Sepsis
Brief Title: Randomized Trial of Inhaled Nitric Oxide to Augment Tissue Perfusion in Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Dr. Trzeciak, PI, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K23GM083211 (NIH); 1K23GM083211-01 (NIH)
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-06

CONDITIONS: Sepsis
Keywords: Sepsis; Severe sepsis; Septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Subjects receive inhaled nitric oxide (40 parts per million) for six hours.
  Interventions: Drug: Inhaled nitric oxide
- 2 (Sham Comparator): Subjects receive sham inhaled nitric oxide for six hours.
  Interventions: Other: Sham inhaled nitric oxide

INTERVENTIONS:
Drug: Inhaled nitric oxide — Inhaled nitric oxide, 40 parts per million, for six hours.
  Other Names: INOmax
  Arms: 1
Other: Sham inhaled nitric oxide — Sham inhaled nitric oxide administration, 0 parts per million, for six hours.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether inhaled nitric oxide is an effective treatment for microcirculatory dysfunction and acute organ system failure in the early stage of sepsis therapy.

DETAILED DESCRIPTION:
Sepsis is a common and devastating disease that is responsible for 215,000 deaths annually in the United States and is the leading cause of death in critically ill patients. Sepsis is now recognized as a time-sensitive emergency, as patients stand the best chance for survival when effective therapeutic interventions are delivered as early as possible. Early goal-directed therapy (EGDT), a protocol-directed resuscitation strategy targeting early optimization of global hemodynamic parameters, can save lives. Use of an EGDT protocol has been associated with the largest mortality benefit demonstrated in sepsis randomized controlled trials to date; however, sepsis still carries an extremely high mortality rate (~30%), even with effective EGDT. As tissue perfusion in sepsis can remain markedly impaired despite normalization of global hemodynamics, targeting macrocirculatory goals of resuscitation (e.g. blood pressure, cardiac output) alone may not be sufficient.

Microcirculatory dysfunction is a pivotal element in the pathogenesis of sepsis. Microcirculatory dysfunction causes impairment of tissue perfusion independent of global hemodynamics, and is hypothesized to be a critical factor in the development of sepsis-induced organ dysfunction, especially in the earliest phase of sepsis therapy. Orthogonal polarization spectral (OPS) videomicroscopy is a technique that permits non-invasive assessment of the microcirculation in human subjects. Using the OPS technique, increasing severity of early microcirculatory derangements in sepsis patients have been associated with acute multi-organ failure and mortality. We recently demonstrated that early derangements of microcirculatory flow in sepsis patients were more severe in non-survivors compared to survivors, even with the application of EGDT. Early recognition of microcirculatory dysfunction and its reversal may lead to improved outcome. Currently, however, there are no therapies to specifically target the microcirculation in sepsis. Novel strategies that go beyond optimization of global hemodynamics and aim to improve microcirculatory blood flow could be a new frontier for sepsis resuscitation. Since the early resuscitation phase of therapy represents the greatest opportunity for impact on clinical outcome in sepsis, it also appears to be the most promising window of opportunity to demonstrate a benefit when investigating novel therapies.

Nitric oxide (NO) is an endogenous molecule that is essential for maintaining microcirculatory homeostasis. Nitric oxide becomes especially critical for protecting microcirculatory patency, integrity, and function when the microcirculation sustains a severe insult (e.g. sepsis). Although NO production is globally upregulated in sepsis, the production of NO is heterogeneous between and within organ systems at the microcirculatory level. We believe that exogenous NO administration may preserve microcirculatory flow in sepsis, and we hypothesize that this will be an effective therapy to augment tissue perfusion. Inhaled nitric oxide (iNO) can deliver NO effectively to the distal microcirculation and "open" low-flow microcirculatory units via modulation of microvascular tone as well as anti-adhesive effects on the microvascular endothelium. Because iNO would not be expected to induce or exacerbate arterial hypotension in sepsis patients, iNO administration is an ideal method to test hypotheses about the effects of exogenous NO on the microcirculation in sepsis.

We hypothesize that iNO will augment microcirculatory perfusion in sepsis resuscitation, and this increase in microcirculatory flow will be associated with improved lactate clearance (an important marker of resuscitation effectiveness) and decreased organ failure (a critical patient-oriented outcome measure). To test our hypothesis, we generated two inter-related specific aims:

Specific Aim 1: To determine whether iNO can augment tissue perfusion in sepsis resuscitation. In a randomized double-blind placebo-controlled trial, we will evaluate the effect of iNO compared to placebo on microcirculatory perfusion indices in sepsis patients who exhibit persistent microcirculatory flow impairment after achievement of global hemodynamic endpoints of resuscitation during EGDT.

Specific Aim 2: To determine whether iNO-mediated improvement in microcirculatory perfusion in sepsis leads to more effective resuscitation and a reduction in organ failure. In a randomized double-blind placebo-controlled trial, we will evaluate the effect of iNO on clinical outcomes of sepsis patients: [(a) increase in lactate clearance from 0-2 hours, and (b) decrease in the Sequential Organ Failure Assessment (SOFA) score from 0 to 24 hours].

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed or suspected infection (acute)

   PLUS:
2. One or both of the following criteria for potential tissue hypoperfusion:

(2a) systolic blood pressure <90 mmHg despite 30cc/kg intravenous crystalloid challenge, OR (2b) serum lactate >4 mmol/L.

Exclusion Criteria:

1. age < 14 years
2. pregnancy
3. "Do Not Resuscitate" status (prior to enrollment)
4. active clinically significant bleeding of any etiology
5. status-post cardiac arrest
6. need for immediate surgery
7. inability to place a sublingual videomicroscopy probe under the tongue (e.g. inability to open the mouth or patient requirement of a high-flow face mask for supplemental oxygen [although videomicroscopy can be performed in patients with an endotracheal tube or nasal cannula])
8. >24 hours elapsed since first documented evidence of meeting criteria for potential tissue hypoperfusion (2a or 2b above).
9. inability to obtain written informed consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Trzeciak, MD, MPH, Principal Investigator — UMDNJ-Robert Wood Johnson Medical School at Camden, Cooper University Hospital, Camden, New Jersey
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

REFERENCES:
- [Background] Trzeciak S, Dellinger RP, Parrillo JE, Guglielmi M, Bajaj J, Abate NL, Arnold RC, Colilla S, Zanotti S, Hollenberg SM; Microcirculatory Alterations in Resuscitation and Shock Investigators. Early microcirculatory perfusion derangements in patients with severe sepsis and septic shock: relationship to hemodynamics, oxygen transport, and survival. Ann Emerg Med. 2007 Jan;49(1):88-98, 98.e1-2. doi: 10.1016/j.annemergmed.2006.08.021. Epub 2006 Nov 7. PMID 17095120
- [Background] Sakr Y, Dubois MJ, De Backer D, Creteur J, Vincent JL. Persistent microcirculatory alterations are associated with organ failure and death in patients with septic shock. Crit Care Med. 2004 Sep;32(9):1825-31. doi: 10.1097/01.ccm.0000138558.16257.3f. PMID 15343008
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Derived] Trzeciak S, Glaspey LJ, Dellinger RP, Durflinger P, Anderson K, Dezfulian C, Roberts BW, Chansky ME, Parrillo JE, Hollenberg SM. Randomized controlled trial of inhaled nitric oxide for the treatment of microcirculatory dysfunction in patients with sepsis*. Crit Care Med. 2014 Dec;42(12):2482-92. doi: 10.1097/CCM.0000000000000549. PMID 25080051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled septic patients in the Emergency Department and Intensive Care Unit
Groups:
- Inhaled Nitric Oxide: Subjects receive inhaled nitric oxide (40 parts per million) for six hours.
- Sham (Comparator): Subjects receive sham inhaled nitric oxide for six hours.
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide | Sham (Comparator)
Started | 26 | 23
Completed | 24 | 22
Not Completed | 2 | 1
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide | Sham (Comparator) | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 14 | 31
  >=65 years | 9 | 9 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (15) | 58 (20) | 58 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  United States | 26 | 23 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in the Sequential Organ Failure Assessment (SOFA) Score
Time Frame: 0-24 hours from protocol initiation
Reporting Status: Not Posted

2. Primary Outcome: Change in Sublingual Microcirculatory Flow Index (MFI)
Description: The MFI is a continuous scale from 0-3, with 3.0 being better outcome and 0.0 being worse outcome.
Time Frame: 0-2 hours of study drug administration
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Inhaled Nitric Oxide | Sham (Comparator)
Number analyzed (Participants) | 24 | 22
units on a scale | -0.06 [-0.19 to 0.04] | -0.03 [-0.13 to 0.17]
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide vs Sham (Comparator); Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.03

3. Secondary Outcome: Lactate Clearance (Blood)
Time Frame: 0-2 hours of study drug administration
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of hospital stay, an average of 5 weeks.
Arm/Group | Inhaled Nitric Oxide | Sham (Comparator)
Serious Adverse Events (participants affected / at risk) | 9/26 | 6/23
Other Adverse Events (participants affected / at risk) | 9/26 | 6/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Nitric Oxide (N=26) | Sham (Comparator) (N=23)
Death (General disorders) | 9 | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Nitric Oxide (N=26) | Sham (Comparator) (N=23)
Death (General disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes